CLINICAL TRIAL: NCT03316417
Title: Adverse Renal Effects of Immune Checkpoints Inhibitors (Nivolumab, Pembrolizumab, Atezolizumab and Ipilimumab) in Clinical Practice: a Large Monocentric Prospective Study
Brief Title: Study of Adverse Renal Effects of Immune Checkpoints Inhibitors
Acronym: ImmuNoTox(INT)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0475
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Adverse Effect; Renal Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients under immunotherapy: All patients with Immune Checkpoints inhibitors treatment (Nivolumab, Pembrolizumab, ipilimumab, Atezolizumab), for dermatologic, pneumologic, or oncologic cancer treated on Centre Hospitalier Lyon Sud are included.
  Interventions: Other: Renal Tolerance to Immunotherapy

INTERVENTIONS:
Other: Renal Tolerance to Immunotherapy — The main objective is to describe the renal tolerance of these innovative therapies within a population homogeneous of patients.

SUMMARY:
Renal toxic events related to Immune Checkpoints Inhibitors therapy (Nivolumab, Pembrolizumab, Atezolizumab and Ipilimumab) have been recently reported. These were immune-allergic acute interstitial nephritis.

However, no systematic study has ever focused on renal adverse effects. The investigators study here the evolution of renal function and the occurrence of nephrological events in a large monocentric cohort of patients treated with Immune Checkpoints Inhibitors in the Centre Hospitalier Lyon Sud. Nephrological parameters based on Serum Creatinine (SCr), estimate Glomerular Filtration Rate (eGFR) and urinary sediment are monitored. The aim of the study is to determine the incidence of renal events due to Immune Checkpoint Inhibitor treatment, particularly Acute Kidney Injury, (AKI) and identify the clinical presentation, histological description and risk factors.

ELIGIBILITY:
Inclusion Criteria:

All patients treated by one of the Immune Checkpoints inhibitors (Nivolumab, Pembrolizumab, ipilimumab or Atezolizumab), for neoplastic pathology in dermatologic, pneumologic, or medical oncology department.

Exclusion Criteria:

* Minor patients (less than 18y).
* Refusal to consent.
* For statistical analysis: Acute Renal Failure caused by another identified etiology than drug toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with Immune Checkpoints inhibitors treatment (Nivolumab, Pembrolizumab, ipilimumab, Atezolizumab), for dermatologic, pneumologic, or oncologic cancer treated on Centre Hospitalier Lyon Sud are included.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute kidney Injury | maximum 6 months
  Acute kidney Injury is defined by the KDIGO (Kidney Disease: Improving Global Outcomes) recommendations by an increase in serum creatinine during follow-up of at least 1.5 times the baseline.
  Follow-up : Nephrological parameters will be notice during whole treatment duration, until interruption for medical reason (tumoral progression, severe adverse event) or end of the study (stop of the collection and analysis of the results); In this case, a 6-month follow-up period for patients undergoing treatment at the time of the collection of data.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No